CLINICAL TRIAL: NCT04421495
Title: Safety and Effectiveness of Delamanid-containing Regimen for Treatment of Patients With Multidrug-resistant Tuberculosis in China
Brief Title: Safety and Effectiveness of Delamanid-containing Regimen for MDR-TB Patients in China
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Chest Hospital (Other)
Responsible Party: Principal Investigator, Liang Li, Vice president, Beijing Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCSY-TB-2020-002
Record Dates: First submitted 2020-06-01; First posted 2020-06-09 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Multidrug Resistant Tuberculosis
Keywords: safety; Delamanid; effectiveness
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant | interventions — OPC-67683

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- delamanid containing regimen arm (Experimental): the only one arm to be studied with delamid-containing regimen.
  Interventions: Drug: Delamanid

INTERVENTIONS:
Drug: Delamanid — the eligible patients will be give damanid-containing regimen
  Other Names: anti-TB new drug containing regimen

SUMMARY:
The purpose of this study is to monitor and evaluate the safety and effectiveness of Delamanid in combination with an optimal background regimen (OBR) of anti-TB drugs for treatment of MDR-TB.

DETAILED DESCRIPTION:
This is a single-arm, multicenter, phase #, open-label trial to evaluate the safety and effectiveness of delamanid-containing regimen in men and women aged 18 to 65 years with microbiologically confirmed pulmonary MDR-TB in China. A target of 600 participants will be enrolled. The study will consist of a screening phase of up to 8 weeks, an open-label study treatment phase of 13-20 months, and a follow-up phase of 12-month after end of study treatment. During the study treatment phase, participants will receive an MDR-TB regimen consisting of 24 weeks of delamanid in combination with 13-20 months of a background regimen.

Participants will be instructed to take their assigned dose of delamanid with at least 3 additional probably effective background drugs according to national and international guidelines. Delamanid dosage will be 100 mg twice daily (b.i.d.) for 24 weeks.

Safety evaluations will include monitoring of AEs, visual acuity testing, routine blood examinations (such as hematology, clinical chemistry, HIV, TSH [for subjects receiving PTO] measurements), urinalysis, and electrocardiograms (ECGs). Participants will initiate treatment with the study regimen if they meet the study eligibility criteria.The end of study will be considered as the last contact for the last participant in the study.

A participant will be considered to have completed the study if he or she has completed the 13-20 months study treatment phase and the required post-treatment follow-up phase. Participants who prematurely discontinue study treatment (unless they withdraw consent) will be followed up for 12 months after end of delamanid treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with microbiologically confirmed multidrug-resistant/rifampicin resistant tuberculosis ;
2. Age 18 to 65 years old;
3. MDR-TB treatment has not been started, or treatment has been started but treatment regimen need to be intensified;
4. According to the guidelines of WHO's consolidated guidelines for the treatment of drug-resistant TB and the consensus of Chinese experts in the treatment of multidrug-resistant and rifampicin resistant TB (2019 edition), effective treatment regimens can only be formed by adding Delamanid based on the results of drug susceptibility testing and the previous treatment history;
5. No history of respiratory failure, no history of cardiac dysfunction and clinically significant arrhythmia, QTcF < 450ms;
6. Patients should be able to take medicines and clinical monitoring according to the requirements of the trial during the treatment and follow-up phases, and adverse effects should be reported to the responsible doctor timely ;
7. Patients should sign the informed consent.

Exclusion Criteria:

1. A history of allergy to nitroimidazole and pyrrole drugs such as Delamanid, metronidazole, tinidazole, or any excipient.
2. Serum transaminase increased ≥3 times the upper limit of normal value or total bilirubin increased ≥2.5 times the upper limit of normal, serum albumin <2.8 g / dL, severe renal impairment.
3. Taking strong CYP3A4 inducer drugs (such as carbamazepine).
4. Is known to be pregnant (or planning to become pregnant) .
5. Participants took part in trials of other new unlisted drugs within the past three months;
6. Congenital QT interval prolongation is known or has any disease that may prolong the QT interval or QTc no less than 500 ms;
7. A history of symptomatic arrhythmia or suffering from clinically related bradycardia;
8. Any cardiac disease that can induce arrhythmias, such as severe hypertension, left ventricular hypertrophy (including hypertrophic cardiomyopathy), or congestive heart failure with reduced left ventricular ejection fraction;
9. Electrolyte disturbance, especially hypokalemia, hypocalcemia or hypomagnesemia;
10. Taking drugs known to prolong the QT interval such as the following drugs (but not limited to) :

    ① Anti-arrhythmic drugs, such as amiodarone, disopyramide, dofetilide, ibutilide, procainamide, quinidine, hydroquinidine, sotalol, etc .;
    * Antipsychotic drugs, such as phenothiazine, sertindole, sultopride, chlorpromazine, haloperidol, mesoridazine, pimozide or thioridazine, and antidepressants; ③ Certain antibiotics, including:

      * Macrolides, such as erythromycin, clarithromycin, etc ;
      * Moxifloxacin, Sparfloxacin;
      * Triazole antifungal drugs;
      * Spray him with amidine;
      * Saquinavir;

        ④ Some non-sedative antihistamines, such as terfenadine, astemizole, mizolastine, etc.
11. Other drugs with protential cardiac risk : cisapride, haloperidol, domperidone, bepridil, diphemanil, probucol, dimepheptanol, methadone, vinblastine, arsenic trioxide.

Deletion criteria:

1. Those who are found to have exclusion items after enrolled;
2. Serious adverse reactions caused by Delamanid, such as allergic reactions, mental disorders, and liver injury (transaminases increase greater than 3 times the upper limit of normal value or total bilirubin increase greater than 2.5 times the upper limit of normal);
3. QTcF ≥500ms or clinically significant ventricular arrhythmia is confirmed;
4. The expert group made decision that it is not appropriate for the patient to continue the treatment with Delamanid;
5. The patient cannot tolerate the background treatment regimen, or the modified background treatment regimen cannot meet the 3 definitive sensitive drugs or 4 probably sensitive drugs;
6. The patient requests dropout.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 608 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2024-07-16 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants experiencing all-cause mortality | from enrollment to the completion of the trial ,an average of 30-32months
  the percentage of participants who died during the trial.
Proportion of participants experiencing treatment-emergent AEs | the whole treatment phase,an average of 18-20 months
  the percentage of participants who experienced adverse effect during treatment phase.

SECONDARY OUTCOMES:
The Percentage of Participants With Sputum Culture Conversion | up to 24 weeks after enrollment
  Sputum culture conversion is defined as 2 consecutive sputum cultures negative for multidrug-resistant tuberculosis (MDR-TB) taken at least 25 days apart.
The Median Time to Sputum Culture Conversion | upto 24 weeks after enrollment
  Sputum culture conversion is defined as 2 consecutive sputum cultures negative for multidrug-resistant tuberculosis (MDR-TB) taken at least 25 days apart.

CONTACTS AND LOCATIONS:
Overall Officials: Liang Li, Principal Investigator — Beijing Chest Hospital
Locations (25):
- China (25):
  - Beijing Chest Hospital, Capital Medical University, Beijing
  - Changsha Central Hospital, Changsha
  - Public Health Clinical Center of Chengdu, Chengdu
  - Chongqing Infectious Disease Medical Center, Chongqing
  - Fuzhou Pulmonary Hospital of Fujian, Fuzhou
  - Guangzhou Chest Hospital, Guangzhou
  - Guiyang Public Health Clinical Center, Guiyang
  - Heilongjiang Province center for tuberculosis Control and Prevention, Haerbin
  - Hangzhou Red Cross Hospital, Hangzhou
  - Jiamusi Tumor Hospital, Jiamusi
  - Tuberculosis Hospital in Jilin Province, Jilin
  - Shandong Provincial Chest Hospital, Jinan
  - The Third People's Hospital of Kunming City, Kunming
  - Lanzhou Pulmonary Hospital, Lanzhou
  - Longtan Hospital of Guangxi Zhuang Autonomous Region, Liuchow
  - Jiangxi Chest (Third People) Hospital, Nanchang
  - Shanghai Pulmonary Hospital, Shanghai
  - Hebei Chest Hospital, Shijiangzhuang
  - The Fifth People Hospital of Suzhou, Suzhou
  - The Fourth People's Hospital of Taiyuan, Taiyuan
  - Wuhan Institute For Tuberculosis Control, Wuhan
  - Wuhan Jinyintan Hospital, Wuhan
  - Shanxi Provincial Tuberculosis Institute, Xi'an
  - Xi'an Chest Hospital, Xi'an
  - Henan Provincial Chest Hospital, Zhengzhou

REFERENCES:
- [Derived] Qin Y, Chen Y, Cai Q. Interim efficacy and safety analysis of the regimen containing delamanid in the treatment of multidrug resistant/rifampicin-resistant/extensively drug-resistant tuberculosis: a single-arm, prospective, monocentric, observational study. BMC Infect Dis. 2025 Dec 19. doi: 10.1186/s12879-025-11945-9. Online ahead of print. PMID 41419836
- [Derived] Yang F, Yin M, Jiang X, Zhao X, An X, Liu Y, Yuan Y. Delamanid-containing regimens over 24 weeks for the treatment of multidrug-resistant/rifampicin-resistant tuberculosis: preliminary results from a single center in a multicenter, prospective, observational study. Front Med (Lausanne). 2025 Sep 29;12:1631030. doi: 10.3389/fmed.2025.1631030. eCollection 2025. PMID 41090140